CLINICAL TRIAL: NCT02914951
Title: Cognitive-Behavioral Therapy for Disruptive Behavior in Children and Adolescents (An Open Pilot Study in Autism Spectrum Disorder)
Brief Title: Cognitive-Behavioral Therapy for Irritability in Children With Autism Spectrum Disorder and Intellectual Disability
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0102012121-D; No NIH funding (Other: 11.14.23)
Record Dates: First submitted 2016-09-20; First posted 2016-09-26 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Autism; Intellectual Disability
Keywords: Autism; Irritability; Disruptive Behavior; Aggression; Behavior Therapy; Cognitive Behavioral Therapy; Intellectual Disability; Cognitive Impairment
MeSH Terms: conditions — Autistic Disorder; Intellectual Disability; Problem Behavior; Aggression; Cognitive Dysfunction | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Behavior therapy for irritability and disruptive behavior for children with autism and intellectual disability
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cognitive-Behavioral Therapy (Experimental): CBT is a behavioral intervention where children are taught various skills for coping with frustration and parents are taught various strategies for managing situations that can be anger-provoking for their child.
  Interventions: Behavioral: Cognitive-Behavioral Therapy; Other: Functional magnetic resonance imaging (fMRI)

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy — CBT is a behavioral intervention that consists of 12 60- to 90-minute-long weekly sessions. A modified, principles-based form of CBT will be used in this study to reduce complexity of activities during therapy sessions while retaining all key elements and principles of CBT.
Other: Functional magnetic resonance imaging (fMRI) — Functional magnetic resonance imaging (fMRI). There will be two fMRI visits, 60 to 90 minute each, one before and the other after CBT. fMRI is a technique that uses magnetism to measure activity of the brain as participants perform simple tasks such as pressing the button in response to pictures. During this study, children will be asked to look at pictures of objects and press or not press the button in response to specific instruction. Participants will also look at pictures of faces and light-point displays depicted biological motion. fMRI is used as an outcome measure to explore if change in irritability is associated with change in brain responses to these tasks during fMRI.

SUMMARY:
In addition to the core symptoms, children and adolescents with Autism Spectrum Disorder (ASD) often exhibit disruptive behavior problems including irritability, tantrums, noncompliance, and aggression. The purpose of this study is to investigate cognitive-behavioral therapy (CBT) for disruptive behavior in children with autism spectrum disorders and intellectual disability. This pilot study will include children with ASD and IQ between 55 and 85 in an open study of CBT. CBT is modified in this study to reduce complexity of activities during therapy sessions but retains all key elements and principles of CBT. Assessments of irritability and disruptive behavior will include clinical interviews, parent ratings and child self-report measures. Study participants will be asked to complete functional magnetic resonance imaging (fMRI) to evaluate biomarkers of social perception and emotion regulation before and after CBT.

DETAILED DESCRIPTION:
Children with ASD share common symptoms in the core domains of social reciprocity, communication, and repetitive behaviors. In addition to the core symptoms, 50 to 70 percent of children with ASD often exhibit disruptive behavior problems including irritability, tantrums, noncompliance, aggression and self-injury.

In this open pilot study expands clinical research on CBT for irritability to children with autism and mild cognitive impairment. CBT consists of individual weekly sessions dedicated to teaching children to recognize situations that may lead to frustration and to build coping skills for dealing with frustration in socially appropriate ways. Recent research as well as clinical reports suggest that children with mild intellectual disabilities (IQ between 55 and 85) can also benefit from CBT. The intervention is modified to reduce complexity of activities during therapy sessions but retains key elements and principles of CBT. Thus, the modified version of CBT is referred to as "Principles-Based Cognitive Behavior Therapy for Irritability in Autism" or PB-CBT for short. Subjects in this study will receive a comprehensive evaluation of ASD and associated psychopathology. Irritability and related disruptive behaviors will be rated on weekly basis to utilize a single-subject approach to data analysis. Children will be asked to participate in functional magnetic resonance imaging (fMRI) with tasks of social perception and emotion regulation before and after CBT. The purpose of the fMRI portion of the study is to evaluate feasibility of fMRI as an outcome measure in studies of behavioral interventions for children with ASD and intellectual disability.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of Autism Spectrum Disorder
* Presence of disruptive behaviors such as irritability and anger outbursts
* IQ between 55 and 85
* ABC Irritability Scale score greater than or equal to 15
* Un-medicated or on stable medication regimen
* Able to complete all study assessment and fMRI procedures

Exclusion Criteria:

* Medical or psychiatric condition that would require alternative treatment

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Estimated)
Dates: Start 2016-10; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Modified Overt Aggression Scale (MOAS) | Weekly - up to 20 weeks
  Modified Overt Aggression Scale (MOAS) is a 16-item scale that reflects the frequency and severity of incidents of aggressive behavior
Aberrant Behavior Checklist - Irritability Scale (ABC-I) | Weekly - up to 20 weeks
  The ABC-I is a 15-item parent rating of irritability that has been commonly used in clinical trials in children with ASD.

SECONDARY OUTCOMES:
Home Situations Questionnaire (HSQ) | baseline
  HSQ is a parent-rated measure of noncompliance in children with ASD
Home Situations Questionnaire (HSQ) | endpoint (16 weeks)
  HSQ is a parent-rated measure of noncompliance in children with ASD

OTHER OUTCOMES:
BOLD signal change in the conditions of the emotion-induction GoNoGo task complete during fMRI scan | baseline
  Participants will perform an emotion-induction GoNoGo task during fMRI
BOLD signal change in the conditions of the emotion-induction GoNoGo task complete during fMRI scan | endpoint (16 weeks)
  Participants will perform an emotion-induction GoNoGo task during fMRI
BOLD signal change during the emotional face perception task completed during fMRI scan | baseline
  Children will perform a task of emotional face perception during fMRI
BOLD signal change during the emotional face perception task completed during fMRI scan | endpoint (16 weeks)
  Children will perform a task of emotional face perception during fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Denis Sukhodolsky, PhD, Principal Investigator — Associate Professor
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States

REFERENCES:
- [Result] Sukhodolsky DG, Smith SD, McCauley SA, Ibrahim K, Piasecka JB. Behavioral Interventions for Anger, Irritability, and Aggression in Children and Adolescents. J Child Adolesc Psychopharmacol. 2016 Feb;26(1):58-64. doi: 10.1089/cap.2015.0120. Epub 2016 Jan 8. PMID 26745682
- [Result] Sukhodolsky DG, Vander Wyk BC, Eilbott JA, McCauley SA, Ibrahim K, Crowley MJ, Pelphrey KA. Neural Mechanisms of Cognitive-Behavioral Therapy for Aggression in Children and Adolescents: Design of a Randomized Controlled Trial Within the National Institute for Mental Health Research Domain Criteria Construct of Frustrative Non-Reward. J Child Adolesc Psychopharmacol. 2016 Feb;26(1):38-48. doi: 10.1089/cap.2015.0164. Epub 2016 Jan 19. PMID 26784537
- See also: Behavior therapy studies for children with autism spectrum disorder at Sukhodolsky lab — https://medicine.yale.edu/lab/sukhodolsky/research/